CLINICAL TRIAL: NCT01765192
Title: A Phase 2, Randomized, Double-Blind, 4-week Crossover Trial to Investigate the Effect of a Once-Daily Combination of 500 µg Roflumilast Plus 10 mg Montelukast vs 10 mg Montelukast Alone on Pulmonary Function, Asthma Symptoms, and Inflammatory Markers in Subjects With Severe Asthma Not Adequately Controlled With a Combination of at Least Medium Dose Inhaled Corticosteroids and Long-Acting Beta Agonists Maintenance Therapy
Brief Title: Roflumilast Plus Montelukast in Adults With Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROF-ASTHMA_202; U1111-1132-3160 (Other: UTN (WHO)); 2012-002064-27 (EudraCT Number); DOH-27-0213-4118 (Registry Identifier: SANCTR)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Drug therapy
MeSH Terms: conditions — Asthma | interventions — Roflumilast; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast plus montelukast, then placebo plus montelukast (Experimental): Participants in sequence 1 received roflumilast 500 μg plus montelukast 10 mg orally once daily for 4 weeks followed by a 4-week washout period and then received placebo plus montelukast 10 mg orally once daily for 4 weeks.
  Interventions: Drug: Roflumilast; Drug: Roflumilast placebo; Drug: Montelukast
- Placebo plus montelukast, then roflumilast plus montelukast (Experimental): Participants in sequence 2 received placebo plus montelukast 10 mg orally once daily for 4 weeks followed by a 4-week washout period and then received roflumilast 500 μg plus montelukast 10 mg orally once daily for 4 weeks.
  Interventions: Drug: Roflumilast; Drug: Roflumilast placebo; Drug: Montelukast

INTERVENTIONS:
Drug: Roflumilast — Roflumilast was supplied in tablets.
  Other Names: Daxas; Daliresp
Drug: Roflumilast placebo — Roflumilast placebo was supplied in tablets.
Drug: Montelukast — Montelukast was supplied in tablets.
  Other Names: Singulair; Pluralair

SUMMARY:
This study will evaluate the effect of roflumilast 500 μg once daily (QD) plus montelukast 10 mg QD versus 10 mg montelukast QD alone on predose (trough) prebronchodilator forced expiratory volume in the first second (FEV1).

DETAILED DESCRIPTION:
The drug being tested in this study is called roflumilast. Roflumilast is being tested to treat people who have asthma. This study will look at lung function and asthma symptoms of people who take roflumilast in combination with montelukast.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements (ie, to follow clinical trial procedures and Investigator instructions adequately).
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a documented physician diagnosis of severe asthma consistent with global initiative for asthma (GINA) step 4 clinical features [Gina 2011] for at least 6 months.
4. Is male or female and aged 18 years or above.
5. Has been treated with a fixed or free combination of at least medium-dose inhaled corticosteroid (ICS) (ie, ≥ 250 µg fluticasone propionate daily or equivalent ICS) plus long-acting beta agonist (LABA) for at least 3 months prior to Screening with stable ICS dose for at least 4 weeks before Visit 2.
6. Shows GINA-defined uncontrolled asthma or an asthma control questionnaire (ACQ-7) score ≥1.5 despite at least medium dose ICS/LABA therapy within 4 weeks prior to Visit 1 (Screening).
7. Shows a pre-bronchodilator FEV1 of > 55% and ≤ 85% of predicted at Visit 1 (Screening). For participants performing induced sputum FEV1 must be in addition > 1 liter.
8. Has airway obstruction proven to be reversible by an improvement of FEV1 of at least 12% and 200 mL after inhalation of a short-acting bronchodilator. This can be either documented in the medical history (with supporting spirometry recordings) in the previous 12 months or demonstrated during screening at Visit 1 (Screening).

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the start of the clinical trial or has participated in the active treatment phase of another clinical trial where a persisting pharmacodynamic effect of the trial treatment of that clinical trial cannot be excluded (eg, participant is well into a treatment free follow-up phase).
2. Participation in another clinical trial during the current trial.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Severe asthma exacerbation not resolved 4 weeks prior to Visit 1, (defined by the need for oral or parenteral glucocorticosteroid intake for at least 3 days and/or hospitalization or emergency room visit with the need for oral or parenteral corticosteroid use).
5. Lower respiratory tract infection not resolved 4 weeks prior to Visit 1.
6. A diagnosis of chronic obstructive pulmonary disease (COPD) (based on Global Initiative for Chronic Obstructive Lung Disease [GOLD] criteria) and/or other relevant forms of lung disease (eg, history of primary bronchiectasis, cystic fibrosis, idiopathic (pan)bronchiolitis or bronchiolitis obliterans, bronchopulmonary allergic aspergillosis, Churg-Strauss Syndrome, paradoxical vocal cord closure, lung resection, lung cancer, interstitial lung disease [eg, fibrosis, silicosis, sarcoidosis], or active tuberculosis) that may interfere with the evaluation of a treatment response.
7. Current participation in a pulmonary rehabilitation program or completion of a pulmonary rehabilitation program within 3 months preceding Visit 1.
8. Has, in the judgment of the investigator, clinically significant abnormal laboratory values (hematology or biochemistry) at screening suggesting an undiagnosed disease requiring further clinical evaluation.
9. Has severe neuropsychiatric or neurological disorders (eg, history of depression associated with suicidal thinking, suicidal ideation or behavior).
10. Has congestive heart failure severity grade III or IV according to the New York Heart Association.
11. Has symptomatic ischemic heart disease (angina pectoris).
12. Has hemodynamically significant cardiac arrhythmias or heart valve deformations.
13. Has liver impairment, defined as Child-Pugh B/C and/or active viral hepatitis.
14. Has severe immunological diseases (eg, multiple sclerosis, systemic lupus erythematosus, progressive multifocal leukoencephalopathy) or known infection with human immunodeficiency virus (HIV).
15. Has severe acute infectious diseases (eg, tuberculosis, or acute hepatitis).
16. Has any diagnosis of a malignant disease (other than basal or squamous cell carcinoma) within 5 years prior to Screening Visit 1.
17. Has a history of smoking within 1 year of Visit 1 and smoking history ≥10 pack years.
18. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day) within the past 1 year prior to the Screening visit.
19. Has history of clinically significant allergies or idiosyncrasies to roflumilast, montelukast or any inactive ingredient(s) of these products, eg, rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, glucose-galactose malabsorption or phenylketonuria.
20. Has known highly unstable asthma defined by severe bronchoconstriction after bronchoprovocation with isotonic saline.
21. Females of childbearing potential not willing to use acceptable contraceptive methods such as hormonal contraceptives (oral, injection or implant) or intrauterine contraceptive devices or who started such methods less than 2 months prior to screening or who are not willing to use a double barrier method of contraception (diaphragm plus condom).
22. If female, is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
23. Is required to take excluded medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (13):
- Germany (6):
  - Berlin
  - Großhansdorf
  - Hamburg
  - Hanover
  - Mainz
  - Schwerin
- Hungary (4):
  - Budapest
  - Nyíregyháza
  - Szarvas
  - Törökbálint
- South Africa (3):
  - Bloemfontein
  - Cape Town
  - Pretoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in Germany, Hungary, and South Africa from 15 February 2013 to 24 October 2013.
Pre-assignment Details: Participants with a historical diagnosis of severe asthma who were inadequately controlled while receiving a combination of at least medium dose inhaled corticosteroids and long-acting beta agonists maintenance therapy were enrolled in 1 of 2 treatment sequences, 500 µg roflumilast plus 10 mg montelukast once daily (QD) or 10 mg montelukast QD.
Period: Treatment Period 1
Arm/Group | Roflumilast Plus Montelukast, Then Placebo Plus Montelukast | Placebo Plus Montelukast, Then Roflumilast Plus Montelukast
Started | 32 | 32
Completed | 32 | 31
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout Period
Arm/Group | Roflumilast Plus Montelukast, Then Placebo Plus Montelukast | Placebo Plus Montelukast, Then Roflumilast Plus Montelukast
Started | 32 | 31
Completed | 30 | 30
Not Completed | 2 | 1
Not completed — Voluntary Withdrawal | 1 | 1
Not completed — Reason not specified | 1 | 0
Period: Treatment Period 2
Arm/Group | Roflumilast Plus Montelukast, Then Placebo Plus Montelukast | Placebo Plus Montelukast, Then Roflumilast Plus Montelukast
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2
Not completed — Reason not specified | 0 | 2
Period: End of Treatment Period 2 to Final Visit
Arm/Group | Roflumilast Plus Montelukast, Then Placebo Plus Montelukast | Placebo Plus Montelukast, Then Roflumilast Plus Montelukast
Started | 30 | 28
Completed | 30 | 27
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set: All randomized participants, analyzed according to the randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Plus Montelukast, Then Placebo Plus Montelukast | Placebo Plus Montelukast, Then Roflumilast Plus Montelukast | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (13.80) | 50.0 (14.10) | 50.1 (13.84)
Age, Customized [Number; unit: participants]
  < 65 years | 27 | 27 | 54
  ≥ 65 years | 5 | 5 | 10
Gender [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 11 | 12 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 0 | 3
  White | 29 | 32 | 61
Region of Enrollment [Number; unit: participants]
  South Africa | 16 | 11 | 27
  Germany | 8 | 12 | 20
  Hungary | 8 | 9 | 17
Height [Mean (Standard Deviation); unit: cm] | 163.7 (8.47) | 168.3 (10.68) | 166.0 (9.85)
Weight [Mean (Standard Deviation); unit: kg] | 79.06 (18.708) | 85.16 (17.491) | 82.11 (18.227)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.53 (7.105) | 30.06 (5.605) | 29.79 (6.354)
Smoking History [Number; unit: participants]
  Never smoked | 22 | 21 | 43
  Current smoker | 0 | 0 | 0
  Ex-smoker | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-Dose (Trough) Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 will be measured using spirometry in accordance with the American Thoracic Society / European Respiratory Society (ATS/ERS) consensus guidelines. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline FEV1 measurement as the covariate was used for analysis.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: Full analysis set: All randomized participants, analyzed according to the randomized treatment with FEV1 data available for analysis after 4 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- Roflumilast Plus Montelukast: Participants received roflumilast 500 μg plus montelukast 10 mg orally once daily for 4 weeks.
- Placebo Plus Montelukast: Participants received placebo plus montelukast 10 mg orally once daily for 4 weeks.
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 58 | 61
liters | 0.18 (0.028) | 0.08 (0.027)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; The primary endpoint was analyzed using an analysis of covariance model adapted for the crossover design. The following fixed factors and covariates were included in the model: Treatment, sequence, period, and baseline FEV1 measurement of the respective treatment period. The reported analysis results are for the 2 crossover treatment periods combined; Test type: Superiority or Other; p = 0.013, ANCOVA; Least Squares (LS) Mean Difference = 0.10, 95% CI 2-sided [0.0219 to 0.1795], Standard Error of Mean 0.039

2. Secondary Outcome: Change From Baseline in Pre-Dose (Trough) Pre-Bronchodilator Forced Vital Capacity (FVC)
Description: FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC will be measured using spirometry in accordance with ATS/ERS consensus guidelines. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline FVC measurement as the covariate was used for analysis.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: Full analysis set: All randomized participants, analyzed according to the randomized treatment with FVC data available for analysis after 4 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 58 | 61
liters | 0.12 (0.029) | 0.06 (0.027)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; Test type: Superiority or Other; p = 0.129, ANCOVA — P-values were obtained using an ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline pre-bronchodilator FVC measurement as the covariate; LS Mean Difference = 0.06, 95% CI 2-sided [-0.0185 to 0.1422], Standard Error of Mean 0.040

3. Secondary Outcome: Change From Baseline in Pre-Dose (Trough) Pre-Bronchodilator Forced Expiratory Flow (FEF) 25-75%
Description: FEF is a measure of how much air can be exhaled from the lungs. It is an indicator of obstruction of the smaller airways. FEF25-75% is the mid-flow rate or forced expiratory flow occurring in the middle 50% of the patient's exhaled volume, and will be measured using spirometry in accordance with ATS/ERS consensus guidelines. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline FEF measurement as the covariate was used for analysis.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: Full analysis set: All randomized participants, analyzed according to the randomized treatment with FEF data available for analysis after 4 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 54 | 55
liters/second | 0.23 (0.039) | 0.11 (0.039)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; Test type: Superiority or Other; p = 0.032, ANCOVA — P-values were obtained using an ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline pre-bronchodilator FEF measurement as the covariate; LS Mean Difference = 0.12, 95% CI 2-sided [0.0113 to 0.2364], Standard Error of Mean 0.056

4. Secondary Outcome: Change From Baseline in Pre-Dose (Trough) Pre-Bronchodilator Peak Expiratory Flow (PEF)
Description: PEF is a person's maximum speed of expiration. It measures the airflow through the bronchi and thus the degree of obstruction in the airways. PEF will be measured using spirometry in accordance with ATS/ERS consensus guidelines. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline PEF measurement as the covariate was used for analysis.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: Full analysis set: All randomized participants, analyzed according to the randomized treatment with PEF data available for analysis after 4 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: liters/minute (L/min)
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 58 | 61
liters/minute (L/min) | 15.05 (10.616) | 7.85 (10.401)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; Test type: Superiority or Other; p = 0.635, ANCOVA — P-values were obtained using an ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline pre-bronchodilator PEF measurement as the covariate; LS Mean Difference = 7.21, 95% CI [-23.0531 to 37.4660], Standard Error of Mean 15.105

5. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF)
Description: PEF will be measured at home using portable electronic peak flow meter. The participant will record PEF daily in the morning immediately after getting up. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline PEF measurement as the covariate was used for analysis.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 60 | 61
L/min | 20.85 (3.708) | 7.23 (3.646)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; Test type: Superiority or Other; p = 0.011, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = 13.62, 95% CI 2-sided [3.1896 to 24.0553], Standard Error of Mean 5.206

6. Secondary Outcome: Change From Baseline in Daytime Asthma Symptoms
Description: Patients will assess their daily day-time asthma symptoms according to the following scale: 0: Very well, no symptoms. 1: One episode of wheezing, cough or breathlessness. 2: More than one episode of wheezing, cough or breathlessness without interfering with normal activities. 3: Wheezing, cough or short of breath most of the day which interfered to some extent with normal activities. 4: Asthma very bad. Unable to carry out daily activities as usual. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline Daytime Asthma Symptoms measurement as the covariate was used for analysis. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: Full analysis set: All randomized participants, analyzed according to the randomized treatment with data available for analysis after 4 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 60 | 61
units on a scale | -0.39 (0.061) | -0.18 (0.063)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; Test type: Superiority or Other; p = 0.025, ANCOVA — P-values were obtained using an ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline Daytime Asthma Symptom Score as the covariate; LS Mean Difference = -0.21, 95% CI 2-sided [-0.3850 to -0.0271], Standard Error of Mean 0.089

7. Secondary Outcome: Change From Baseline in Nighttime Asthma Symptoms
Description: Patients will assess their daily night-time asthma symptoms according to the following scale: 0: No symptoms, slept through the night. 1: Slept well but some complaints in the morning. 2: Woke up once because of asthma (inclusive early awakening). 3: Woke up several times because of asthma (inclusive early awakening). 4: Bad night, awake most of the night because of asthma. An ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline Nighttime Asthma Symptoms measurement as the covariate was used for analysis. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Days 1 and 56) and after 4 weeks of treatment (Days 28 and 84)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Number analyzed (Participants) | 60 | 61
units on a scale | -0.27 (0.053) | -0.17 (0.052)
Statistical Analysis 1: Comparison: Roflumilast Plus Montelukast vs Placebo Plus Montelukast; Test type: Superiority or Other; p = 0.217, ANCOVA — P-values were obtained using an ANCOVA model with treatment sequence, treatment period, and study treatment as fixed factors with Baseline Nighttime Asthma Symptoms measurement as the covariate; LS Mean Difference = -0.09, 95% CI 2-sided [-0.2426 to 0.0563], Standard Error of Mean 0.075

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Days 1-105)
Description: Safety analysis set: All randomized participants who received at least 1 dose of study drug. Adverse events are reported for 61 and 62 participants in the roflumilast + montelukast (R+M) and placebo + montelukast (P+M) groups, respectively, as 3 participants discontinued prior to receiving R+M and 2 participants discontinued prior to receiving P+M.
Arm/Group | Roflumilast Plus Montelukast | Placebo Plus Montelukast
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 5/61 | 0/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Plus Montelukast (N=61) | Placebo Plus Montelukast (N=62)
Headache (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.